CLINICAL TRIAL: NCT01064921
Title: A Phase I Trial Of Vorinostat In The Treatment Of Advanced Laryngeal, Hypopharyngeal, Nasopharyngeal And Oropharyngeal Squamous Cell Carcinoma Of The Head And Neck.
Brief Title: Ph I Vorinostat in the Treatment of Advanced Staged Oropharyngeal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Matthew Old, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09120; NCI-2009-01606 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx
Keywords: oropharyngeal cancer; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms | interventions — Vorinostat; Cisplatin; Radiotherapy; Radiation; Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat on days 0-2 and cisplatin IV on days 7, 21 and 35. Patients undergo radiation therapy 5 days a week beginning on day 7. Patients also receive concurrent oral vorinostat along with the radiotherapy to be given 3 days per week (Monday, Tuesday, and Wednesday). Optional repeat tumor and normal mucosal biopsies will be performed and blood will be drawn for correlative studies.
  Interventions: Drug: vorinostat; Drug: cisplatin; Radiation: radiation therapy; Procedure: Correlative Studies

INTERVENTIONS:
Drug: vorinostat — The first vorinostat dose level is 100mg, and the second dose will be 200mg, third dose will be 300mg. If the first vorinostat dose level is found to be excessively toxic, the patient will be reduced to -1 dosing level then if still too toxic reduced again to dose level -2. Dose escalation of vorinostat will continue in increments of 100 mg (i.e., 200 mg on dosing days, 300 mg on dosing days). Vorinostat will be given 3 consecutive days per week (e.g. Monday, Tuesday, Wednesday).
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin; PDD
Radiation: radiation therapy — Standard chemoradiation therapy X 7 weeks (Days 7-56), concurrent with oral Vorinostat given three days per week (Mon, Tues, Wed)
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: Correlative Studies — Day 35, 2 weeks post radiation therapy completion optional tumor/normal muscosal biopsy and blood draw for correlative studies. At day 153 an optional tumor/normal tissue biopsy and blood draw for correlative studies.
  Other Names: blood draw; biopsy

SUMMARY:
RATIONALE: Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Giving vorinostat together with chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat when given together with cisplatin and radiation therapy in treating patients with stage III or stage IVa squamous cell cancer of the oropharynx which is either unresectable or borderline resectable.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose of Vorinostat in combination with concurrent chemoradiotherapy for the treatment of advance stage OPSCC.

SECONDARY OBJECTIVES:

l. To determine the complete response rate, overall survival and progression free survival using the maximally tolerated dose of Vorinostat.

TERTIARY OBJECTIVES:

I. To assess treatment related acute and late toxicities when combining Vorinostat with chemoradiation and correlate these toxicities to molecular markers of apoptosis in tumor and normal oral mucosa.

II. To evaluate the effect of Vorinostat on tumor immune surveillance, particularly in HPV positive patients.

III. To illustrate that Vorinostat alters the methylation status of commonly methylated genes in OPSCC.

OUTLINE: This is a dose-escalation study of vorinostat. Patients receive oral vorinostat on days 0-2 and cisplatin IV on days 7, 21, and 35. Patients undergo radiotherapy 5 days a week beginning on day 7. Patients also receive concurrent oral vorinostat along with the radiotherapy to be given 3 days per week (Monday, Tuesday, and Wednesday). Treatment continues for 7 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed unresectable or borderline resectable squamous cell carcinoma of the oropharynx will be eligible for enrollment to the clinical trial
* Oropharyngeal sites of tumor include tonsil, soft palate, base of tongue, lateral and posterior pharyngeal wall
* Patient must be AJCC (American Joint Committee on Cancer) Stage III (T3N0, T1-2N1) or Stage IVa (T1-4N2-3M0, T4N0-1 M0) and be either unresectable or borderline resectable
* No prior therapy for the tumor, including extensive surgery, radiation therapy, chemotherapy, immunotherapy, targeted therapy or any other investigational agents; surgical biopsy prior to beginning the study is allowable
* Prior malignancies at sites other than the head and neck are allowable if there has been greater than or equal to a 3 year disease free interval; basal cell carcinoma of the skin and in-situ cervix dysplasias are allowable within this 3 year interval if completely resected
* There must be documentation of evaluable tumor within four weeks of beginning therapy
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0-2, (Karnofsky > 60%)
* Ability to understand and the willingness to sign a written informed consent
* Patient must have normal liver and bone marrow function
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin Time or INR (international normalized ratio) =< 1.5x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* K levels preferred normal limits with no clinical abnormalities
* Mg levels preferred normal limits with no clinical abnormalities
* Creatinine =< ULN OR Calculated creatinine clearance >= 50 mL/min
* Serum total bilirubin =< 1.5 X ULN
* AST (SGOT) and ALT (SGPT) =< 2.5 X ULN
* Alkaline Phosphatase =< 2.5 X ULN
* No known malabsorption syndrome
* Female patients of childbearing potential must be willing to use birth control; the 2 birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy, used throughout the study starting with visit 1
* The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner) or sponge; other methods of contraception such as copper intrauterine device or spermicide may be used
* Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents); female patient of childbearing potential has a negative serum pregnancy test β-hCG within 7 days prior to receiving the first dose of vorinostat
* Male patients agree to use an adequate method of contraception for the duration of the study
* The patient must have a life expectancy of at least 12 weeks
* Patients on coumadin therapy are eligible for study

Exclusion Criteria:

* Major surgery or trauma occurring within 28 days of starting the trial
* History of allergic reactions attributed to compounds similar in chemical or biological composition to Vorinostat or other agents used in this study
* Gastrointestinal tract disease or previous surgical procedures resulting in an inability to take oral or enteral medication or a requirement for IV alimentation
* Pregnant women; breast feeding should be discontinued during treatment
* Active peptic ulcer disease
* Uncontrolled comorbid illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina, untreated or new cardiac arrhythmia, psychiatric or social condition which would limit the patient's understanding of and compliance with the study
* Prisoners and other vulnerable populations
* Patients who have had prior treatment with an HDAC inhibitor (e.g., romidepsin (Depsipeptide), NSC-630176, MS 275, LAQ-824, belinostat (PXD-101), LBH589, MGCD0103, CRA024781, etc)
* Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug(s)
* Patients with known active viral hepatitis or known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat in combination with concurrent chemoradiation therapy | Weekly during treatment; Every 2 weeks for the first month after treatment completion; Then every 4 weeks until day 153
The toxic effects of the combination of vorinostat and cisplatin using NCI CTCAE v. 4.0 | Weekly during treatment; Every 2 weeks for the first month after treatment completion; Then every 4 weeks until day 153

SECONDARY OUTCOMES:
Tumor responses to vorinostat or vorinostat combined with chemoradiation. | Days 35, 56 then after Day 153 every 12 weeks for 24 months
Complete response rate | Days 35, 56 then after Day 153 every 12 weeks for 24 months
Overall survival | Days 35, 56 then after Day 153 every 12 weeks for 24 months
Progression free survival | Days 35, 56 then after Day 153 every 12 weeks for 24 months
Relationship between Vorinostat therapy and tumor suppressor genes product assessed by Fas and FasL protein expression level in tumor and the normal mucosa | Before, post SAHA treatment, and post the concurrent chemoradiation /SAHA therapy
HPV-specific T-cell in patients with HPV+ tumors | After the run in period of vorinostat but before the start of RT; Day 35; 2 weeks after the completion of RT; Day 153

CONTACTS AND LOCATIONS:
Overall Officials: Old Matthew, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu